CLINICAL TRIAL: NCT03966378
Title: Reminerlization Potential of Grape Seeds Extract Gel Versus Casein Phosphopeptide-amorphous Calcium Phosphate in Carious White Spot Lesions in Post Orthodontic Patients
Brief Title: Reminerlization Potential of GSE Gel versusCPP-ACP in Carious White Spot Lesions in Post Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aseel Saleh Omeran, pricipal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 607
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — amorphous calcium phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grape seeds extract (Experimental): Every week the grape seeds extract (gel) put into the tray and apply it to the upper teeth of the participant.
  Interventions: Other: Grape seeds extract
- Casein-phosphopeptide/amorphous-calcium phosphate (Active Comparator): CPP-ACP paste apply to the teeth twice daily.
  Interventions: Other: Casein-phosphopeptide/amorphous-calcium phosphate

INTERVENTIONS:
Other: Grape seeds extract — Grape seeds extract powder
  Arms: Grape seeds extract
Other: Casein-phosphopeptide/amorphous-calcium phosphate — CPP-ACP paste
  Arms: Casein-phosphopeptide/amorphous-calcium phosphate

SUMMARY:
Assess the effectiveness of applying grape seed extract (GSE) gel versus casein phosphopeptide-amorphous calcium phosphate (MI) paste on remineralization of white spot lesion (WSLs) in post orthodontic patients.

DETAILED DESCRIPTION:
The development of WSLs is a challenging problem in the track of orthodontic treatment. Especially in patients wearing fixed orthodontic appliances, plaque accumulation increases around brackets and bands and the pH on dental surfaces becomes acidic.

These early lesions are willing to remineralization, arrest, reharden and revert to healthy enamel condition through a remineralization process involving the diffusion of minerals into the defective tooth structure. For this purpose various remineralizing agents such as casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) and grape seed extract (GSE) have been used.

This research is conducted for early intervention and treatment of the white spot lesions by non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two WSLs on the labial surfaces of six maxillary anterior teeth that were not present before orthodontic therapy.

Exclusion Criteria:

* Severe or active periodontal disease.
* Patients had received therapeutic irradiation to the head and neck region.
* Patients had participated in a clinical trial within 6 months before commencement of this trial.
* Patients unable to return for recall appointments
* Presence of abnormal oral, medical, or mental condition (including any milk-related allergies or any medical condition involving kidneys or salivary glands).
* Presence of restorations or cavities in any anterior teeth or enamel hypoplasia, dental fluorosis, or intrinsic and extrinsic pigmentation.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-03 (Estimated); Primary Completion 2020-04-06 (Estimated); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
Quantitative changes of white spot lesions | evaluation of tooth surface changes at baseline and at 4, 12, and 24 weeks after starting treatment .
  changes in fluorescence of white spot lesions will be evaluated after reminerlization by using diagnodent device by score (0-20).